CLINICAL TRIAL: NCT00808821
Title: Pharyngeal Carriage Rates and Genetic Typing of Group A Streptococcus and Streptococcus Pneumonia Among Israeli Military Basic Trainees
Status: Completed | Type: Observational
Sponsor: Medical Corps, Israel Defense Force (Other)
Other Study IDs: 544-2006-IDF-CTIL
Record Dates: First submitted 2008-12-15; First posted 2008-12-16 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-10

CONDITIONS: Carriage; Group A Streptococcus; Streptococcus Pneumonia
MeSH Terms: conditions — Pneumonia

SUMMARY:
The study is aimed at assessing pharyngeal and nasopharyngeal Streptococcus pneumonia carriage and pharyngeal Group A streptococcus carriage among field units new recruits.

ELIGIBILITY:
Inclusion Criteria:

* Israeli Military Basic Trainee

Exclusion Criteria:

* None

Age Groups: Child, Adult, Older Adult